CLINICAL TRIAL: NCT07004738
Title: Ultrasound Assessment of Rectus Abdominis Muscle Thickness and Residual Bladder Volume Before and After Pelvic Floor Exercises
Brief Title: Assessment of Rectus Abdominis Muscle Thickness and Residual Bladder Volume Before and After Pelvic Floor Exercises
Acronym: Ultrasound
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7377
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pelvic Floor Disorders
Keywords: pelvic floor exercises; rectus abdominis muscle thickness; residual bladder
MeSH Terms: conditions — Pelvic Floor Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor exercise group (Experimental): Participants will be instructed to perform daily pelvic floor exercises under the guidance of a physical therapist specializing in pelvic health. The exercises focus on isolated pelvic muscle contractions and core muscle engagement. The exercises will be performed 3 times per day for 6 weeks.
  Interventions: Other: Pelvic floor exercises
- Control Group (Other): Women in this group who have been diagnosed with pelvic floor dysfunction will not be given any exercises. Women will continue their routine lives and their evaluations will be made.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Pelvic floor exercises — The bladder should be emptied before the exercise. In order to correctly identify the pelvic floor muscles, it is necessary to initially try to hold urine while emptying the bladder. If the result is successful, it means that the correct muscles have contracted. During the learning phase, the exercise can be done in a supine position with the legs bent at the knees or in a sitting position. Initially, the pelvic floor muscles should be contracted for 5 seconds by pulling them inward as if stopping the passage of urine or gas, and then rested for 5 seconds.
  Arms: Pelvic floor exercise group
Other: Control group — Women in this group who have been diagnosed with pelvic floor dysfunction will not be given any exercises. Women will continue their routine lives and their evaluations will be made.
  Arms: Control Group

SUMMARY:
The study will be conducted on 40 women between the ages of 20-40 who volunteer to participate in the study. All participants will be selected from individuals who have been diagnosed with pelvic floor dysfunction and have no history of pelvic surgery. Pelvic floor dysfunction will be diagnosed by an Obstetrics and Gynecology Specialist. Participants will be divided into two groups as the Pelvic floor exercise group and the control group.

DETAILED DESCRIPTION:
The study will be conducted on 40 women between the ages of 20-40 who volunteer to participate in the study. All participants will be selected from individuals who have been diagnosed with pelvic floor dysfunction and have no history of pelvic surgery. Pelvic floor dysfunction will be diagnosed by an Obstetrics and Gynecology Specialist. Participants will be divided into two groups as the Pelvic floor exercise group and the control group. Group distributions will be made by randomization.org website. Participants in the pelvic floor exercise group will be instructed to do daily pelvic floor exercises under the guidance of a physiotherapist specialized in pelvic health. No exercises will be given to women diagnosed with pelvic floor dysfunction in this group. Women will continue their routine lives and their evaluations will be made.

ELIGIBILITY:
Inclusion Criteria:

* were being between 20-40 years of age,
* having pelvic floor dysfunction,
* not having any problems that would prevent performing pelvic floor exercises

Exclusion Criteria:

* previous pelvic surgery
* active urinary tract infections
* neurological conditions affecting bladder control

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The gender eligibility is based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Measurements | 20 minutes
  Ultrasound measurements will be performed at two points: at baseline (before the exercise program) and after 6 weeks of intervention. A high-resolution ultrasound device will be used to measure the thickness and cross-sectional area of the rectus abdominis muscle at rest.
The residual bladder volume measurement | 20 minutes
  The residual bladder volume immediately after voiding will also be measured by ultrasonography to assess bladder control.A normal post-void residual volume is between 50 mL (milliliters) and 100 mL.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, Assoc. Prof., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will be shared where necessary.

REFERENCES:
- [Result] Wang X, Li H, Luan B, Han R, Lun W. Dynamic Evaluation of the Rectus Abdominis Muscle before and after Delivery by Ultrasonography. Evid Based Complement Alternat Med. 2022 Aug 26;2022:9751136. doi: 10.1155/2022/9751136. eCollection 2022. PMID 36062170
- See also: Dynamic Evaluation of the Rectus Abdominis Muscle before and after Delivery by Ultrasonography — https://pubmed.ncbi.nlm.nih.gov/36062170/